CLINICAL TRIAL: NCT01752140
Title: A Prospective Randomized Trial of Prostate Biopsy Protocols Comparing the Vienna Nomogram and a Standard 10-core Biopsy Scheme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Santa Maria, Portugal (Other)
Responsible Party: Principal Investigator, Tito Palmela Leitão, Dr., Hospital de Santa Maria, Portugal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BPTRVienna
Record Dates: First submitted 2012-12-13; First posted 2012-12-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Prostate biopsy; Vienna nomogram
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10-core prostate biopsy protocol group (Active Comparator): Ultrasound guided prostate biopsy with extraction of 10 cores
  Interventions: Procedure: 10-core prostate biopsy protocol
- Vienna nomogram prostate biopsy protocol group (Active Comparator): Ultrasound guided prostate biopsy performed according to the Vienna nomogram
  Interventions: Procedure: Vienna nomogram prostate biopsy protocol

INTERVENTIONS:
Procedure: 10-core prostate biopsy protocol — Local vascular bundle anesthesia with 2% lidocaine was performed using a 22G Chiba needle. Ultrasound guided prostate biopsy using a standard biopsy device to obtain 10 biopsy cores.
  Arms: 10-core prostate biopsy protocol group
Procedure: Vienna nomogram prostate biopsy protocol — Local vascular bundle anesthesia with 2% lidocaine was performed using a 22G Chiba needle. Ultrasound guided prostate biopsy using a standard biopsy device to obtain a number of cores as defined by the Vienna nomogram.
  Arms: Vienna nomogram prostate biopsy protocol group

SUMMARY:
In this study, the investigators aim to determine if the Vienna nomogram increases the detection rate of TRUS-guided prostate biopsies by conducting a prospective randomized study comparing the Vienna nomogram with a 10-core biopsy protocol.

DETAILED DESCRIPTION:
Trans rectal ultrasound (TRUS) guided prostate biopsy remains the standard for prostate cancer diagnosis. However, the standard protocols miss 15 to 30% of cancers, leading to a variable number of repeat biopsies.

In 2005 the Vienna nomogram was introduced, defining the number of cores to be obtained in a prostate biopsy in relation to age and prostate volume in patients with a serum PSA level of 2-10 ng/mL.

The objective of the study is to determine if the Vienna nomogram increases the detection rate of trans rectal ultrasound guided prostate biopsies, compared to a 10-core biopsy.

This prospective randomized study enrolled men eligible for a prostate biopsy were randomized to a Vienna nomogram protocol or a 10-core protocol. They were further stratified according to age (≤65; >65 and ≤70; >70 years) and prostate volume (≤30; >30 and ≤50; >50 and ≤70; >70 cc).

A subgroup analysis for patients with serum PSA values between 2 and 10 ng/mL was performed.

ELIGIBILITY:
Inclusion Criteria:

* PSA elevation
* Abnormal digital rectal examination
* Abnormal findings on prostate imaging

Exclusion Criteria:

* Active urinary tract infection
* Documented previous pathological prostatitis
* History of urinary retention
* Recent lower urinary tract surgery

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Prostate cancer detection rate | Up to four weeks after intervention

SECONDARY OUTCOMES:
Prostate cancer detection rate in prostate volume and age subclasses | Up to four weeks after intervention
Gleason score concordance between biopsy and prostatectomy specimens | Up to four weeks after prostatectomy

CONTACTS AND LOCATIONS:
Overall Officials: Tito P Leitão, Dr., Principal Investigator — Hospital de Santa Maria
Locations (1):
- Urology Department - Hospital de Santa Maria, Lisbon, Lisbon District, Portugal

REFERENCES:
- [Background] Uzzo RG, Wei JT, Waldbaum RS, Perlmutter AP, Byrne JC, Vaughan ED Jr. The influence of prostate size on cancer detection. Urology. 1995 Dec;46(6):831-6. doi: 10.1016/s0090-4295(99)80353-7. PMID 7502425
- [Background] Djavan B, Margreiter M. Biopsy standards for detection of prostate cancer. World J Urol. 2007 Mar;25(1):11-7. doi: 10.1007/s00345-007-0151-1. Epub 2007 Mar 7. PMID 17342490
- [Background] Lecuona A, Heyns CF. A prospective, randomized trial comparing the Vienna nomogram to an eight-core prostate biopsy protocol. BJU Int. 2011 Jul;108(2):204-8. doi: 10.1111/j.1464-410X.2010.09887.x. Epub 2010 Nov 19. PMID 21087452
- [Background] Remzi M, Fong YK, Dobrovits M, Anagnostou T, Seitz C, Waldert M, Harik M, Marihart S, Marberger M, Djavan B. The Vienna nomogram: validation of a novel biopsy strategy defining the optimal number of cores based on patient age and total prostate volume. J Urol. 2005 Oct;174(4 Pt 1):1256-60; discussion 1260-1; author reply 1261. doi: 10.1097/01.ju.0000173924.83392.cc. PMID 16145388